CLINICAL TRIAL: NCT05909423
Title: Combining Intratumoral Flu Vaccine and Systemic Pembrolizumab in Patients With Early pMMR Colorectal Cancer - the FLU-IMMUNE Trial.
Brief Title: Combining Intratumoral Flu Vaccine and Systemic Pembrolizumab in Patients With Early pMMR Colorectal Cancer
Acronym: FLU-IMMUNE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: Slagelse Hospital (Other)
Responsible Party: Principal Investigator, Ismail Gögenur, Professor, DMSc, Zealand University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-503228-17-00
Record Dates: First submitted 2023-05-18; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Influenza Vaccines; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): Intratumoral flu vaccine treatment Systemic single dose pembrolizumab treatment
  Interventions: Drug: Influenza vaccine; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Influenza vaccine — Intratumoral influenza vaccine treatment, administered via endoscopic procedure
Drug: Pembrolizumab — Single dose pembrolizumab treatment

SUMMARY:
Immune checkpoint inhibitor (ICI) treatment has produced striking results in patients with colorectal cancer (CRC) of the subtype deficient mismatch repair (dMMR). The majority of patients, however, have proficient MMR (pMMR) tumors, with limited effect of ICIs. The key difference between dMMR and pMMR tumors is the infiltration of cytotoxic T-cells. dMMR tumors have increased infiltration and thus increased efficacy from ICI treatment. The investigators conducted a proof of concept study where the investigators applied an intratumoral (IT) unaltered flu vaccine in ten patients with non-metastatic pMMR CRC. The intervention increased infiltration of cytotoxic T-cells and the immune checkpoint PD-L1, suggesting that IT flu vaccine primes pMMR tumors to ICI treatment. The investigators aim to test the combination of IT flu vaccine and ICI treatment in patients with non-metastatic pMMR CRC in a new trial. The hypothesis is that IT flu vaccine and ICI treatment will synergistically to induce cancer cell death.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically confirmed localized pMMR stage cT1N0M0 to cT4N2M0 (stage I to III) colorectal adenocarcinoma.
* Have indication for elective curative intended surgery without neoadjuvant therapy.
* Be ≥ 18 years of age on the date of signing the informed consent.
* Provide written informed consent
* Have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Have adequate bone marrow function:
* Hemoglobin ≥ 6.2 mmol/L or ≥ 10 g/dL
* Absolute neutrophil count (ANC) ≥ 1.5 × 109/L
* Platelet count ≥ 100 × 109/L
* Have adequate kidney function defined as Glomerular filtration rate (GFR) ≥ 60 mL/min or creatinine ≤1.5 X upper limit of normal (ULN)
* Have adequate liver function defined as:

  * Total bilirubin ≤ 1.5 × ULN
  * Alanine aminotransferase (ALT): ≤ 2.5 × ULN
  * Alkaline phosphatase: ≤ 2.5 × ULN
* Follow the conditions regarding fertility, pregnancy, and lactation:

  o Female and male participants of reproductive potential (for definition refer to appendix 18) must agree to avoid becoming pregnant or impregnating a partner, respectively, while receiving pembrolizumab and for 180 days after the administration.
* Participants must use (or have their partner use) an acceptable method of contraception, as outlined in the appendix 16, during heterosexual activity, while receiving pembrolizumab and for 120 days after the administration.
* Women of reproductive potential (WORP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to receiving pembrolizumab.
* Women must not be breastfeeding.

Exclusion Criteria:

* Has any serious or uncontrolled medical disorder that, in the opinion of the investigator or treating physician, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results.
* Has an autoimmune disorder (except thyroiditis with replacement therapy and type I diabetes mellitus).
* Has received prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody or any other antibody/drug specifically targeting T cell co-stimulation or checkpoint pathways.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies), active chronic or acute Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA is detected).
* Has a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Has received live vaccines within 30 days prior to first dose trial treatment (Examples of live vaccines include, but are not limited to: measles, mumps, rubella, chickenpox,
* Has recently received yellow fever, rabies, BCG, and typhoid (oral) vaccine.
* Has a history of allergy to study drug components or a history of severe hypersensitivity reaction to any monoclonal antibody
* Any previous allergic reaction to influenza vaccine or constituents, egg and chicken proteins, neomycin, formaldehyde or octoxinol-9
* Acute febrile illness
* Acute infectious disease
* Highly inflamed gastrointestinal tissue which is ulcerated and bleeding

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Pathological response | Day 30-35
  The primary endpoint will be the percent of viable tumor cells in the resected specimen. Partial response will be defined as at least 30% tumor regression and major pathological response (MPR) will be defined as < 10 % viable cells corresponding to Mandard tumor regression grade 1-2

SECONDARY OUTCOMES:
Number of participants with specific treatment-related adverse events as assessed by CTCAE v4.0" | Day 0-365
  Intratumoral flu vaccine treatment:
  The specific safety endpoint is perforation at tumor site due to intratumoral flu vaccine treatment
  Pembrolizumab treatment:
  Postponement of surgery, and surgical complication that leads to reoperation
  The Departments of Surgery are responsible for assessment of the "Before pembrolizumab treatment" safety endpoint, while Department of Surgery and Oncology are responsible for assessment of the remaining safety endpoints. Causality assessment will be done by investigators or delegates with relevant experience by use of the WHO-UMC causality assessment system.
Tumor microenvironment | Day 0-35
  Immunohistochemical analysis of CD3+ and CD8+ T cells, spatial protein expression analyses of immune-infiltrated regions of tumors at the different time points, flow cytometry, and full transcriptomic analyses including single cell analysis.
Analysis of perturbations in the immune activity with a focus on effector and memory CD8+ T cells | Day 0-35
  Flow cytometry and full transcriptomic analyses including single cell analysis of effector and memory CD8+ T cells

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Surgical Science, Department of Surgery, Zealand University Hospital, Koege, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided